CLINICAL TRIAL: NCT00966966
Title: An Open-Label, Nonrandomized Study To Evaluate The Potential Pharmacokinetic Interaction Between SAM-531 and Gemfibrozil, A Cytochrome P-450 2C8 Inhibitor, When Coadministered Orally To Healthy Young Adult Subjects
Brief Title: Study Evaluating Potential Interaction Between SAM-531 And Gemfibrozil When Co-Administered
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3193A1-1109; B1961001
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531; Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SAM-531_gemfibrozil
  Interventions: Drug: SAM-531 and gemfibrozil

INTERVENTIONS:
Drug: SAM-531 and gemfibrozil — 2 single doses of 5 mg SAM-531 (capsules) a daily dose of 1200 mg Gemfibrozil (one tablet of 600mg at approximately 8 a.m. and one tablet of 600 mg at approximately 6 p.m.) for 14 days

SUMMARY:
The purpose of this study is to evaluate the effects of multiple doses of Gemfibrozil on the plasma concentration of a single dose of SAM-531 in healthy young adult subjects and to assess the safety and tolerability of co-administration of SAM-531 and Gemfibrozil.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index in the range of 18 to 30 kg/m2 and body weight greater than 50 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination findings, clinical laboratory test results, vital sign measurements, and digital 12-lead ECG readings.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal (GI), endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 24 days
Time to maximum plasma concentration (tmax) | 24 days
Area under the concentration-time curve (AUC) | 24 days

SECONDARY OUTCOMES:
Safety as measured by adverse event monitoring, ECG, vital signs, and laboratory tests | 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Utrecht, Netherlands

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3193A1-1109&StudyName=Study%20Evaluating%20Potential%20Interaction%20Between%20SAM-531%20And%20Gemfibrozil%20When%20Co-Administered